CLINICAL TRIAL: NCT03541746
Title: The Value of Using Platelet Rich Plasma After Hysteroscopic Lysis of Severe Intrauterine Adhesions (A Randomized Controlled Trial)
Brief Title: The Value of Using Platelet Rich Plasma After Hysteroscopic Lysis of Severe Intrauterine Adhesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Mahmoud Abd El-Wahab Torky, Principal Investigator, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PRP-HLIUA
Record Dates: First submitted 2018-02-13; First posted 2018-05-31 (Actual); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Intrauterine Adhesion
MeSH Terms: conditions — Gynatresia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Platelet Rich Plasma
  Interventions: Biological: Platelet Rich Plasma
- Control Group (Active Comparator): Intrauterine Foley's Catheter
  Interventions: Device: Intrauterine Foley's Catheter

INTERVENTIONS:
Biological: Platelet Rich Plasma — After hysteroscopic adhesiolysis, 30 patients will undergo once injection of 5ml PRP into the wall then lining the uterine cavity by 5ml platelet rich plasma gel. Finally, Foley balloon catheter will be inserted intrauterine then inflated and cutting its stem and to be left for two weeks.
  Arms: Study Group
Device: Intrauterine Foley's Catheter — After hysteroscopic adhesiolysis, 30 patients will undergo intrauterine insertion of one inflated Foley balloon catheter with cutting its stem only to be left for two weeks.
  Arms: Control Group

SUMMARY:
The aim of present study is to evaluate the effect of the use of platelet rich plasma in decreasing recurrence of intrauterine adhesions after its lysis.

DETAILED DESCRIPTION:
Research question:

In women undergoing hysteroscopic adhesiolysis, does postoperative use of platelet rich plasma decrease the recurrence of intrauterine adhesions?

Research hypothesis:

In women undergoing hysteroscopic adhesiolysis for Asherman's syndrome, postoperative use of platelet rich plasma may decrease the recurrence of intrauterine adhesions.

ELIGIBILITY:
Inclusion Criteria:

* Infertility due to Asherman's syndrome with history of hypomenorrhea or amenorrhea and infertility and evaluated by office hysteroscopy to confirm the presence of sever adhesions according to American fertility society.

Exclusion Criteria:

* Hb < 11 g/dL, platelets < 150.000/mm3
* Patient taking anticoagulant.
* Patient taking NSAID in the 10 days before procedure.
* Any significant comorbidity or psychiatric disorder that would compromise patient's consent.
* Active cervical or uterine infection.

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Prevent recurrence of intrauterine adhesions | Reassessed after one month
  Prevent recurrence of intrauterine adhesions after hysteroscopic adhesiolysis assessed by office hysteroscopy according to American Fertility Society adhesion score:
  1. Extent of cavity involved: ( <1/3, 1/3 - 2/3, >2/3 )
  2. Type of adhesions: (filmy, filmy to dense, dense)
  3. menstrual pattern (normal, hypomenorrhea, amenorrhea)

SECONDARY OUTCOMES:
Return of menses | Reassessed after one month
  Return/normalization of expected menses by history (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed I Amer, MD, Study Chair — Professor; Mortada E Ahmed, MD, Study Director — Lecturer; Reda M Kamal, MD, Study Director — Lecturer
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Egypt